CLINICAL TRIAL: NCT00629876
Title: A Phase 1, Multicenter, Open-Label Dose Escalation Study Evaluating the Safety and Tolerability of Multiple Hematide Injections in Subjects With Refractory Non-Small Cell Lung Cancer, Breast Cancer, or Prostate Cancer Who Are Anemic and Receiving Cytotoxic Chemotherapy
Brief Title: A Safety and Tolerability Study of Peginesatide in Anemic Cancer Patients Receiving Cytotoxic Chemotherapy.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the uncertain regulatory landscape for erythropoiesis-stimulating agents in oncology indications.
Sponsor: Takeda (Industry)
Collaborators: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM_101; U1111-1126-1765 (Registry Identifier: WHO)
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Anemia
Keywords: Chemotherapy; Drug Therapy
MeSH Terms: conditions — Anemia | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginesatide (Experimental)
  Interventions: Drug: Peginesatide

INTERVENTIONS:
Drug: Peginesatide — Peginesatide 0.075, 0.1, 0.125, 0.15, 0.175, 0.2, 0.225 or 0.25 mg/kg administered subcutaneously every 3 weeks for a total of at least 2 doses. Subsequent injections given every 3 weeks thereafter regardless of the schedule of subsequent chemotherapy cycles.
  Following Study Day 43, subjects may continue on Peginesatide treatment, dosing every 3 weeks until 4 weeks after discontinuation of taxane-containing chemotherapy regimen, the occurrence of a dose limiting toxicity, documented disease progression or change in chemotherapy regimen.
  Other Names: Hematide

SUMMARY:
The purpose of this study is to determine the safety and tolerability of peginesatide used to treat anemia in subjects diagnosed with recurrent non-small cell lung cancer, breast cancer or prostate cancer and who also receiving a taxane chemotherapy.

DETAILED DESCRIPTION:
Currently approved erythropoiesis stimulating agents have been used successfully to increase hemoglobin levels, reduce fatigue and other anemia-related symptoms, improve daily function, and alleviate the need for transfusions of red blood cells in subjects with chronic kidney disease-related anemia or in cancer subjects with chemotherapy-induced anemia.

Peginesatide (hematide) Injection is a parenteral formulation for administration by intravenous or subcutaneous injection that is being developed for the correction of anemia in patients with chronic kidney disease, including patients on dialysis and patients not on dialysis, and for the treatment of patients with anemia due to concomitantly administered chemotherapy.

This is a multicenter, open-label dose escalation study to evaluate the safety, tolerability, and efficacy of multiple doses of peginesatide Injection in subjects with refractory non-small cell lung cancer, breast cancer, or prostate cancer. These subjects must have anemia diagnosed as a result of taxane chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Individuals with one of the following histologically confirmed tumors:

  * stage IIIB/IV non-small-cell lung cancer
  * metastatic breast cancer
  * androgen insensitive prostate cancer and are scheduled to receive at least 4 weeks of chemotherapy, including a taxane.
* Has progression or relapse after treatment with at least one regimen of chemotherapy or hormone therapy.
* Has a hemoglobin value of greater than or equal to 8 and less than 10.5 g/dL within 1 week prior to administration of study drug.
* Has an Eastern Cooperative Oncology Group Performance Status of 0-2.
* Has one ferritin level greater than or equal to 100 ng/mL within 4 weeks prior to study drug administration.
* Has one serum or red cell folate level above the lower limit of normal within 4 weeks prior to study drug administration.
* Has one vitamin B12 level above the lower limit of normal within 4 weeks prior to study drug administration.
* Has one absolute neutrophil count greater than or equal to 1.5 x 109/L within 1 week prior to administration of study drug.
* The subject has a serum creatinine less than or equal to 1.5 mg/dL or a measured creatinine clearance greater than 60 mL/min.
* The subject has one platelet count greater than or equal to 100 x 109/L within 1 week prior to administration of study drug.
* The subject has a Life expectancy greater than 4 months.
* The subject has a body mass index between 18 and 30 kg/m2, inclusive, prior to study drug administration.
* The subject has a negative test result for hepatitis B surface antigen, and hepatitis C virus antibody at Screening.

Exclusion Criteria:

* Has a history of failure to respond to erythropoiesis-stimulating agent treatment.
* Has had treatment with any erythropoiesis-stimulating agent in the past 4 weeks.
* Is known to have antibodies to other erythropoiesis-stimulating agents or history of Pure Red Cell Aplasia.
* Has received Peginesatide in a previous clinical study or as a therapeutic agent.
* Has a history of hypersensitivity or allergies to Peginesatide, other erythropoiesis-stimulating agents or related compounds.
* Has had red blood cell transfusion within 4 weeks prior to study drug administration.
* Has known hemoglobinopathy (eg, homozygous sickle-cell disease, thalassemia of all types, etc).
* Has known hemolytic condition.
* Has known blood loss as a cause of anemia, iron deficiency anemia, or anemia caused by gastrointestinal bleeding.
* Has any previous or planned radiotherapy to more than 30% of active bone marrow.
* Has donated more than 400 mL of blood within the 90 days preceding the beginning of the study.
* Has known intolerance to parenteral iron supplementation.
* Has received IV iron within 1 week of study drug administration.
* Has history of bone marrow or peripheral blood cell transplantation.
* Has central nervous system metastases.
* Has a history of deep venous thrombosis, pulmonary embolism or other thrombotic event (eg, stroke, myocardial infarction, etc.) in the previous 6 months or known history of hypercoagulable disorder.
* Has uncontrolled, or symptomatic inflammatory disease (eg, rheumatoid arthritis, systemic lupus erythematosus, etc).
* Has poorly controlled hypertension per the investigator's judgment within 4 weeks prior to study drug administration (eg, systolic greater than or equal to 170 mm Hg or diastolic greater than or equal to 100 mm Hg on repeat readings).
* Has had a seizure in the 6 months prior to study drug administration.
* Has advanced chronic congestive heart failure - New York Heart Association Class III or IV.
* Has a history or presence of an abnormal electrocardiogram at Screening that, in the investigator's opinion, is clinically significant.
* Has a known history of human immunodeficiency virus.
* Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as consumption of more than 4 alcoholic drinks per day) within 1 year prior to Baseline.
* Has aspartate aminotransferase or alanine aminotransferase greater than 2.5 times the upper limit of normal (aspartate aminotransferase or alanine aminotransferase greater than 5 times the upper limit of normal if liver metastases are present), active liver disease or jaundice.
* Is currently taking or anticipated to require anticoagulants other than aspirin (eg, coumadin, ticlopidine, etc.).
* Has a bilirubin greater than the upper limit of normal.
* Has pyrexia/fever greater than or equal to 39°C within 48 hours prior to study drug administration.
* Has high likelihood of early withdrawal or interruption of the study (eg, myocardial infarction within the past 3 months, severe or unstable coronary artery disease, stroke, respiratory, autoimmune, neuropsychiatric or neurological abnormalities, or any other clinically significant medical diseases or conditions within the prior 6 months that may, in the investigator's opinion, interfere with assessment or follow-up of the subject).
* Has anticipated elective surgery during the study period.
* Has exposure to any investigational agent within 1 month prior to administration of study drug or planned receipt during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose. | End of Treatment.

SECONDARY OUTCOMES:
Proportion of subjects who have 2 consecutive Hgb values of either an increase of ≥1 g/dL or a Hgb ≥11 g/dL in the absence of a red blood cell transfusion. | At All Visits for every cycle.
Proportion of subjects who have an increase in Hgb of ≥1 g/dL or a Hgb ≥11 g/dL in the absence of a red blood cell transfusion. | Days 22 and 43 for every cycle.
Proportion of subjects with 2 consecutive Hgb values increase of ≥1 g/dL or ≥11 g/dL during the Treatment phase absent of red blood cell transfusion within the prior 28 days and without excursion of Hgb values above 12 g/dL for ≥2 consecutive weeks. | Within the prior 28 days of every cycle for a minimum of 2 consecutive weeks.
Proportion of subjects who received at least 1 RBC transfusion. | From Day 29 to End of Treatment for every cycle.
Change from Baseline in Hemoglobin. | At Each Visit for every cycle.
Duration of maintaining Hgb values within the range of 10.5 g/dL and 12.0 g/dL. | At Each Visit for every cycle.
Pharmacokinetics of Peginesatide (PK Cohort Only). | At Each Visit for every cycle.
Adverse events and serious adverse events. | At All Visits for every cycle.
Physical examination (including weight, vital signs, and oral temperature). | At All Visits for every cycle.
Clinical Laboratory Tests and Electrocardiograms. | At All Visits for every cycle.
Electrocardiograms. | At Final Visit for every cycle.
Signs and symptoms for thromboembolytic events. | At All Visits for every cycle.
Proportion of subjects who have incidence of Hgb values >12 g/dL. | At All Visits for every cycle.
Proportion of subjects who have Hgb increases by more than 1 g/dL in a 2-week period. | At All Visits for every cycle.
Tumor progression. | Every 2 cycles of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Clinical Science, Study Director — Takeda
Locations (2):
- United States (2):
  - Jacksonville, Florida
  - Corpus Christi, Texas